CLINICAL TRIAL: NCT05823779
Title: A 48 Week Observational Study of the Frequency of Symptomatic Herpes Virus I and II in HIV Infected Subjects
Acronym: HSVHIV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Global Research Institute (Industry)
Collaborators: Rational Vaccines Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: GlobalResearch
Record Dates: First submitted 2023-04-09; First posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: HIV Disease; Herpes Simplex 1; Herpes Simplex 2
Keywords: HIV, Herpes Simplex 1, Herpes Simplex 2
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We are retaining patient serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood draw — We will be drawing blood for verify HIV status, HSV 1 or 2 antibodies, CD4 and HIV-PCR

SUMMARY:
This study is an observational, cohort, prospective study looking at the frequency of Herpes Simplex Virus (HSV) 1 and or 2 outbreaks in HIV positive patients who's HIV virus is controlled on highly active anti-retroviral therapy. We will be enrolling fifty (50) patients.

DETAILED DESCRIPTION:
We will be confirming that the patients are HIV positive and has antibodies to either HSV 1 or HSV 2 as part of the screening process. If so, we will then obtain patient baseline HIV-PCR, CD4, medial history including medications on day one. Whether the patient is on any or no herpes controlling medication. If the patient has what they feel is a flare up of HSV, they will come into clinic where the lesion will be culture and the patient's HIV-PCR and CD4 will also be obtained. Otherwise, the patient will receive phone follow ups every three months to see if there has been and change in their health or medications. The main endpoint is to see if there is a correlation between outbreaks in HIV patients and their CD4 cells and/or HIV and/or Herpes medication.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be 18 years or older at the time of screening
2. Males, Females, Transgender Male and Transgender Females
3. HIV positive
4. Positive antibody to HSV- 1/and or HSV-2
5. If Female of child baring potential, documented negative pregnancy test at the time of screening.

Exclusion Criteria:

1. Active opportunistic infection
2. Current chemotherapy
3. Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are positive for HIV antibodies and IgG or IgM antibodies to Herpes Simplex Virus 1 or Herpes Simplex Virus 2
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Epidemiology | 48 weeks
  The frequency of HSV outbreaks in HIV positive patients.

SECONDARY OUTCOMES:
Co Morbidity | 48 weeks
  Correlation of HSV outbreak with patient CD4 count and/or HIV-PCR

CONTACTS AND LOCATIONS:
Locations (1):
- Global Research Institute, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Share with Rational Vaccine
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: At conclusion of the study
Access Criteria: Total Access